CLINICAL TRIAL: NCT04855175
Title: Evaluation of Cranioplasty Using Native Bone Autograft Versus Synthetic Bone Allograft
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor termination
Sponsor: LifeBridge Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1682010
Record Dates: First submitted 2021-04-09; First posted 2021-04-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Surgical Procedure, Unspecified
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Autograft group (Active Comparator): The autologous group will receive bone harvested from the patient's own body
  Interventions: Other: Autograft
- Allograft group (ClearFit) (Active Comparator): The allograft group will receive a synthetic bone known as ClearFit
  Interventions: Device: Synthetic Bone Allograft (ClearFit)

INTERVENTIONS:
Device: Synthetic Bone Allograft (ClearFit) — Patients in this arm will receive ClearFit (synthetic bone allograft)
  Arms: Allograft group (ClearFit)
Other: Autograft — Patients in this arm will use patient's own bone
  Arms: Autograft group

SUMMARY:
Elevated intracranial pressure (ICP) is a common neurosurgical emergency that may arise from several conditions, which cause an intracranial mass effect. In the case of conservatively refractory ICP elevation, one viable treatment option is ICP-lowering surgery, i.e., decompressive craniectomy (DC) in which a large portion of the skull bone is removed and the dura mater opened, creating more room for the brain tissue to expand and thus reducing the ICP. A successful CP will restore the contour of the cranium, protect the brain, and ensure a natural ICP, and some patients also show neurological improvement post-CP. Thus, CP has a great potential for improving the patient's quality of life.

Bone flap resorption (BFR) implies weakening and loosening of the autologous bone flap after reimplantation and is regarded as a late CP complication involving nonunion of the bone flap with the surrounding bone margins and cavity formation in the flap itself, which eventually necessitates removal of the bone flap and a new CP using a synthetic implant. These additional operations increase costs and necessitate further hospital stays, while rendering the patient vulnerable to additional complications.

Prior research performed as part of the FDA approval process has shown the ASPCI's to be a safe and effective means of performing cranial reconstruction, the anticipated risks do not differ from the risks faced by a patient undergoing either option as they are both currently considered standards of care.

This study will evaluate the overall patient outcomes of cranial reconstruction surgery using native bone autograft as compared to using synthetic bone allograft.

DETAILED DESCRIPTION:
Elevated intracranial pressure (ICP) is a common neurosurgical emergency that may arise from several conditions, which cause an intracranial mass effect. In the case of conservatively refractory ICP elevation, one viable treatment option is ICP-lowering surgery, i.e., decompressive craniectomy (DC) in which a large portion of the skull bone is removed and the dura mater opened, creating more room for the brain tissue to expand and thus reducing the ICP. In many centers, the bone flap removed in DC is customarily kept deep frozen at -70°C until reimplantation during cranioplasty (CP). The cranium is repaired during CP by returning the previously removed autologous bone flap or by placing an artificial implant in the defect area. A successful CP will restore the contour of the cranium, protect the brain, and ensure a natural ICP, and some patients also show neurological improvement post-CP1-4. Thus, CP has a great potential for improving the patient's quality of life. Although widely regarded as a routine operation, CP often involves serious complications, such as postoperative hemorrhages, surgical site infection (SSI), and, most importantly, resorption of the autologous bone flap5-8.

Bone flap resorption (BFR) implies weakening and loosening of the autologous bone flap after reimplantation and is regarded as a late CP complication involving nonunion of the bone flap with the surrounding bone margins and cavity formation in the flap itself, which eventually necessitates removal of the bone flap and a new CP using a synthetic implant. These additional operations increase costs and necessitate further hospital stays, while rendering the patient vulnerable to additional complications. The reported prevalence of BFR with autologous CPs has varied significantly, from 1.4% to 32.0%, with infection rates ranging from 4.6% to 16.4%9-12.

CP is a common procedure for cranial reconstruction in the setting of trauma, stroke, skull neoplasm, osteomyelitis, or after procedures that are approached via craniectomy such as microvascular decompression or acoustic neuroma.

Recently there have been two major areas of interest presenting in the literature. First, there have been at least 6 manuscripts published on retrospective data comparing autologous bone versus synthetic prosthetic for CP13-18. Each has shown benefit for synthetic prosthetics. However, the community is resistant to implement a treatment pattern where synthetic bone is a "first line" choice for CP. Therefore, a prospective randomized controlled trial is needed to understand with high confidence the option that is most beneficial for patients.

Prior research performed as part of the FDA approval process has shown the ASPCI's to be a safe and effective means of performing cranial reconstruction, the anticipated risks do not differ from the risks faced by a patient undergoing either option as they are both currently considered standards of care.

This study will evaluate the overall patient outcomes of cranial reconstruction surgery using native bone autograft as compared to using synthetic bone allograft.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients being considered for CP surgery by the investigating physician at the Life Bridge Health-Sinai Hospital of Baltimore
* Able to read and speak English, or have LAR who reads and speaks English
* Patients who need cranial reconstruction

Exclusion Criteria:

* Patients affected by comminuted skull fractures,
* Patients affected by osteomyelitis,
* Patients with skull neoplasm and therefore not be candidates for autologous CP
* Patients who would need to be allocated to one group over the other due to clinical presentation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
To compare the surgical and post-operative outcomes (complications) of two standard of care cohorts: autograft versus allograft (ClearFit) | intraoperatively
  Asses for infection, hematomas, fractures, mobilization and scar retraction, wound site infection, UTI, pneumonia, delayed internal bleeding, reoperation, and hardware failure
To compare the surgical and post-operative outcomes (complications) of two standard of care cohorts: autograft versus allograft (ClearFit) | post-operatively through study completion, an average of 1 year
  Asses for infection, hematomas, fractures, mobilization and scar retraction, wound site infection, UTI, pneumonia, delayed internal bleeding, reoperation, and hardware failure
To compare the surgical and post-operative outcomes (complications) of two standard of care cohorts: autograft versus allograft (ClearFit) | 2 weeks post-operation
  Asses for infection, hematomas, fractures, mobilization and scar retraction, wound site infection, UTI, pneumonia, delayed internal bleeding, reoperation, and hardware failure
To compare the surgical and post-operative outcomes (complications) of two standard of care cohorts: autograft versus allograft (ClearFit) | 6 weeks post-operation
  Asses for infection, hematomas, fractures, mobilization and scar retraction, wound site infection, UTI, pneumonia, delayed internal bleeding, reoperation, and hardware failure
To compare the surgical and post-operative outcomes (complications) of two standard of care cohorts: autograft versus allograft (ClearFit) | 3 months post-operation
  Asses for infection, hematomas, fractures, mobilization and scar retraction, wound site infection, UTI, pneumonia, delayed internal bleeding, reoperation, and hardware failure
To compare the surgical and post-operative outcomes (complications) of two standard of care cohorts: autograft versus allograft (ClearFit) | 6 months post-operation
  Asses for infection, hematomas, fractures, mobilization and scar retraction, wound site infection, UTI, pneumonia, delayed internal bleeding, reoperation, and hardware failure
To compare the surgical and post-operative outcomes (complications) of two standard of care cohorts: autograft versus allograft (ClearFit) | 1 year post-operation
  Asses for infection, hematomas, fractures, mobilization and scar retraction, wound site infection, UTI, pneumonia, delayed internal bleeding, reoperation, and hardware failure
To assess change in surgical and post-operative outcomes (function) of two standard of care cohorts: autograft versus allograft (ClearFit) | 24 hours post operation, 2 weeks, 6 weeks, 3 months, 6 months, 1-year
  Barthel index consisting of 10 questions - score range 0 (completely dependent)- 20 (completely independent)
To assess change in surgical and post-operative outcomes (function) of two standard of care cohorts: autograft versus allograft (ClearFit) | 24 hours post operation, 2 weeks, 6 weeks, 3 months, 6 months, 1-year
  Karnofsky scale (0-100); 0 indicating death and 100 indicating no additional help is needed
To assess change the surgical and post-operative outcomes (function) of two standard of care cohorts: autograft versus allograft (ClearFit) | 24 hours post operation, 2 weeks, 6 weeks, 3 months, 6 months, 1-year
  Glasgow Outcome Scale (GOS) on a scale of 1(death)- 5 (good recovery)

SECONDARY OUTCOMES:
To assess change in pain using the Visual Analogue Scale (VAS) Pain scale | 24 hours post operation, 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  Assess change in pain; ranking pain on a scale of 1 (least amount of pain)-10 (greatest amount of pain)
To assess change in disability using the Oswestry Disability Index (ODI) | 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  Assess change in disability; 6 item questionnaire; scores range from 0(minimal d disability)-60 (bed bound)
To assess change in quality of life using the Health and Quality of life improvement (SF-36) | 2 weeks, 6 weeks, 3 months, 6 months, and 1 year
  Assess change in quality of life; 36-item questionnaire, 0 (favorable health state life)-100 (poor health state)
To assess overall patient satisfaction of two standard of care cohorts: autograft versus allograft (ClearFit)Patient Satisfaction | at the 2 week visit
  Patient Satisfaction questionnaire; 5 questions; scores range from 0(unsatisfied) - 22(completely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: William Ashley, MD, PhD, MBA, Principal Investigator — Sinai Hospital of Baltimore
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coelho F, Oliveira AM, Paiva WS, Freire FR, Calado VT, Amorim RL, Neville IS, de Andrade AF, Bor-Seng-Shu E, Anghinah R, Teixeira MJ. Comprehensive cognitive and cerebral hemodynamic evaluation after cranioplasty. Neuropsychiatr Dis Treat. 2014 May 2;10:695-701. doi: 10.2147/NDT.S52875. eCollection 2014. PMID 24833902
- [Background] Di Stefano C, Rinaldesi ML, Quinquinio C, Ridolfi C, Vallasciani M, Sturiale C, Piperno R. Neuropsychological changes and cranioplasty: A group analysis. Brain Inj. 2016;30(2):164-71. doi: 10.3109/02699052.2015.1090013. Epub 2015 Dec 8. PMID 26647093
- [Background] Honeybul S, Janzen C, Kruger K, Ho KM. The impact of cranioplasty on neurological function. Br J Neurosurg. 2013 Oct;27(5):636-41. doi: 10.3109/02688697.2013.817532. Epub 2013 Jul 25. PMID 23883370
- [Background] Shahid AH, Mohanty M, Singla N, Mittal BR, Gupta SK. The effect of cranioplasty following decompressive craniectomy on cerebral blood perfusion, neurological, and cognitive outcome. J Neurosurg. 2018 Jan;128(1):229-235. doi: 10.3171/2016.10.JNS16678. Epub 2017 Mar 3. PMID 28298042
- [Background] Stieglitz LH, Fung C, Murek M, Fichtner J, Raabe A, Beck J. What happens to the bone flap? Long-term outcome after reimplantation of cryoconserved bone flaps in a consecutive series of 92 patients. Acta Neurochir (Wien). 2015 Feb;157(2):275-80. doi: 10.1007/s00701-014-2310-7. Epub 2014 Dec 24. PMID 25534126
- [Background] Sundseth J, Sundseth A, Berg-Johnsen J, Sorteberg W, Lindegaard KF. Cranioplasty with autologous cryopreserved bone after decompressive craniectomy: complications and risk factors for developing surgical site infection. Acta Neurochir (Wien). 2014 Apr;156(4):805-11; discussion 811. doi: 10.1007/s00701-013-1992-6. Epub 2014 Feb 4. PMID 24493001
- [Background] Martin KD, Franz B, Kirsch M, Polanski W, von der Hagen M, Schackert G, Sobottka SB. Autologous bone flap cranioplasty following decompressive craniectomy is combined with a high complication rate in pediatric traumatic brain injury patients. Acta Neurochir (Wien). 2014 Apr;156(4):813-24. doi: 10.1007/s00701-014-2021-0. Epub 2014 Feb 16. PMID 24532225
- [Background] Klinger DR, Madden C, Beshay J, White J, Gambrell K, Rickert K. Autologous and acrylic cranioplasty: a review of 10 years and 258 cases. World Neurosurg. 2014 Sep-Oct;82(3-4):e525-30. doi: 10.1016/j.wneu.2013.08.005. Epub 2013 Sep 13. PMID 24036124
- [Background] Moreira-Gonzalez A, Jackson IT, Miyawaki T, Barakat K, DiNick V. Clinical outcome in cranioplasty: critical review in long-term follow-up. J Craniofac Surg. 2003 Mar;14(2):144-53. doi: 10.1097/00001665-200303000-00003. PMID 12621283
- [Background] Chang V, Hartzfeld P, Langlois M, Mahmood A, Seyfried D. Outcomes of cranial repair after craniectomy. J Neurosurg. 2010 May;112(5):1120-4. doi: 10.3171/2009.6.JNS09133. PMID 19612971
- [Background] Walcott BP, Kwon CS, Sheth SA, Fehnel CR, Koffie RM, Asaad WF, Nahed BV, Coumans JV. Predictors of cranioplasty complications in stroke and trauma patients. J Neurosurg. 2013 Apr;118(4):757-62. doi: 10.3171/2013.1.JNS121626. Epub 2013 Feb 8. PMID 23394335
- [Background] Korhonen TK, Tetri S, Huttunen J, Lindgren A, Piitulainen JM, Serlo W, Vallittu PK, Posti JP. Predictors of primary autograft cranioplasty survival and resorption after craniectomy. J Neurosurg. 2018 May 11;130(5):1672-1679. doi: 10.3171/2017.12.JNS172013. Print 2019 May 1. PMID 29749908
- [Background] Malcolm JG, Mahmooth Z, Rindler RS, Allen JW, Grossberg JA, Pradilla G, Ahmad FU. Autologous Cranioplasty is Associated with Increased Reoperation Rate: A Systematic Review and Meta-Analysis. World Neurosurg. 2018 Aug;116:60-68. doi: 10.1016/j.wneu.2018.05.009. Epub 2018 May 16. PMID 29753896
- [Background] van de Vijfeijken SECM, Munker TJAG, Spijker R, Karssemakers LHE, Vandertop WP, Becking AG, Ubbink DT; CranioSafe Group. Autologous Bone Is Inferior to Alloplastic Cranioplasties: Safety of Autograft and Allograft Materials for Cranioplasties, a Systematic Review. World Neurosurg. 2018 Sep;117:443-452.e8. doi: 10.1016/j.wneu.2018.05.193. Epub 2018 Jun 5. PMID 29879511
- [Background] Schoekler B, Trummer M. Prediction parameters of bone flap resorption following cranioplasty with autologous bone. Clin Neurol Neurosurg. 2014 May;120:64-7. doi: 10.1016/j.clineuro.2014.02.014. Epub 2014 Feb 24. PMID 24731578
- [Background] Lethaus B, Bloebaum M, Essers B, ter Laak MP, Steiner T, Kessler P. Patient-specific implants compared with stored bone grafts for patients with interval cranioplasty. J Craniofac Surg. 2014 Jan;25(1):206-9. doi: 10.1097/SCS.0000000000000396. PMID 24406579
- [Background] Pryor LS, Gage E, Langevin CJ, Herrera F, Breithaupt AD, Gordon CR, Afifi AM, Zins JE, Meltzer H, Gosman A, Cohen SR, Holmes R. Review of bone substitutes. Craniomaxillofac Trauma Reconstr. 2009 Oct;2(3):151-60. doi: 10.1055/s-0029-1224777. PMID 22110809
- [Background] Gordon CR, Huang J, Brem H. Neuroplastic Surgery. J Craniofac Surg. 2018 Jan;29(1):4-5. doi: 10.1097/SCS.0000000000004063. No abstract available. PMID 29077688
- [Background] Huang GJ, Zhong S, Susarla SM, Swanson EW, Huang J, Gordon CR. Craniofacial reconstruction with poly(methyl methacrylate) customized cranial implants. J Craniofac Surg. 2015 Jan;26(1):64-70. doi: 10.1097/SCS.0000000000001315. PMID 25376145
- [Background] Zins JE, Moreira-Gonzalez A, Papay FA. Use of calcium-based bone cements in the repair of large, full-thickness cranial defects: a caution. Plast Reconstr Surg. 2007 Oct;120(5):1332-1342. doi: 10.1097/01.prs.0000279557.29134.cd. PMID 17898609
- [Background] Aydin S, Kucukyuruk B, Abuzayed B, Aydin S, Sanus GZ. Cranioplasty: Review of materials and techniques. J Neurosci Rural Pract. 2011 Jul;2(2):162-7. doi: 10.4103/0976-3147.83584. PMID 21897681
- [Background] Ashayeri K, M Jackson E, Huang J, Brem H, Gordon CR. Syndrome of the Trephined: A Systematic Review. Neurosurgery. 2016 Oct;79(4):525-34. doi: 10.1227/NEU.0000000000001366. PMID 27489166
- [Background] Segal DH, Oppenheim JS, Murovic JA. Neurological recovery after cranioplasty. Neurosurgery. 1994 Apr;34(4):729-31; discussion 731. doi: 10.1227/00006123-199404000-00024. PMID 8008174
- [Background] Wolff A, Santiago GF, Belzberg M, Huggins C, Lim M, Weingart J, Anderson W, Coon A, Huang J, Brem H, Gordon C. Adult Cranioplasty Reconstruction With Customized Cranial Implants: Preferred Technique, Timing, and Biomaterials. J Craniofac Surg. 2018 Jun;29(4):887-894. doi: 10.1097/SCS.0000000000004385. PMID 29489570